CLINICAL TRIAL: NCT00527748
Title: The Use of a New Foot and Ankle Range of Motion (Stretching) Apparatus in Subjects With Stiff Ankles
Brief Title: Foot and Ankle Range of Motion (Stretching) Apparatus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left institution. No data analysis completed.
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1092357
Record Dates: First submitted 2007-09-07; First posted 2007-09-11 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-03

CONDITIONS: Plantar Fasciitis; Flatfoot; Calcaneus Fractures
Keywords: Range of Motion; Ankle Fractures; Elderly patients
MeSH Terms: conditions — Fasciitis, Plantar; Flatfoot; Ankle Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of care (No Intervention): Patient ankle range of motion will be assessed at clinic visit. No stretching exercises with the device, but will be provided standard care through physiotherapist in acute cases, and no stretching exercises for chronic patients. Reassessment will be done at six weeks and 10 weeks.
- Non-Measuring Ankle Exerciser (Experimental): Subjects will train using only one combination of movement, dorsiflexion with inversion. This is done by manipulating the ring so that the medial and anterior ropes are taut. Subject will start with 3 minute warm-up. Subject will then manipulate the ring so that the foot moves into dorsiflexion with inversion until a point of tolerable discomfort is felt; subject will hold this position for 30 seconds. Stretch will be repeated 10 times, each day, for six weeks. Reassessment will be done at six weeks and 10 weeks.
  Interventions: Device: Non-Measuring Ankle Exerciser

INTERVENTIONS:
Device: Non-Measuring Ankle Exerciser — Stretching exercise performed 10 times per day, for six (6) weeks.
  Other Names: Ankle Recovery Mechanism (ARM)
  Arms: Non-Measuring Ankle Exerciser

SUMMARY:
Range of motion at ankle joint and subtalar joint will be assessed before and after utilization of ARM device. The changes in range of motion will be recorded and compared to literature.

DETAILED DESCRIPTION:
The purpose of this study is to assess how effective a new device is in increasing range of motion and reducing stiffness in the foot and ankle of patients with acquired flatfoot, patients with plantar fasciitis, and those suffering from stiffness after cast removal or other lengthy immobilization.

Project will utilize a physical therapist to measure range of motion and stiffness when patients are consented. Patients will be re-measured at six weeks following use of the device to assist in stretching ankle and foot muscles, and again at 10 weeks for final stiffness and range of motion assessment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* stiffness in or about the ankle joint due to age, diabetes, trauma, flatfoot, plantar fasciitis, or immobilization

Exclusion Criteria:

* not physically able to use device
* patients with pain disorders
* patients lacking necessary hand-eye coordination
* patients using lower extremity external fixator
* patients with history of non-compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-09; Primary Completion 2011-12 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saul G Trevino, MD, Principal Investigator — University of Missouri-Columbia School of Medicine
Locations (1):
- University of Missouri-Columbia Healthcare, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 26 participants were enrolled. While we know the number who completed the study (23), we do not know to which group/arm they were assigned. There are no other recruitment details, study results or data available as the PI left the institution without making this information available to the research department.
Groups:
- Standard of Care or Ankle Exerciser: Patient ankle range of motion will be assessed at clinic visit. They will either receive standard care physiotherapy, or use the ankle exerciser in the following manner:
  Subjects will train using only one combination of movement, dorsiflexion with inversion. This is done by manipulating the ring so that the medial and anterior ropes are taut. Subject will start with 3 minute warm-up. Subject will then manipulate the ring so that the foot moves into dorsiflexion with inversion until a point of tolerable discomfort is felt; subject will hold this position for 30 seconds. Stretch will be repeated 10 times, each day, for six weeks.
  Reassessment will be done at six weeks and 10 weeks.
Period: Overall Study
Arm/Group | Standard of Care or Ankle Exerciser
Started | 26
Completed | 23
Not Completed | 3
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Population: Although 23 participants completed the study, we do not know their baseline characteristics or to which arm/group they were assigned as the investigator left the institution without making this information available.
Groups:
- Standard of Care or Ankle Exerciser: Patient ankle range of motion will be assessed at clinic visit. They will either receive standard care physiotherapy, or use the ankle exerciser in the following manner:
  Subjects will train using only one combination of movement, dorsiflexion with inversion. This is done by manipulating the ring so that the medial and anterior ropes are taut. Subject will start with 3 minute warm-up. Subject will then manipulate the ring so that the foot moves into dorsiflexion with inversion until a point of tolerable discomfort is felt; subject will hold this position for 30 seconds. Stretch will be repeated 10 times, each day, for six weeks.
  Reassessment will be done at six weeks and 10 weeks.Patient ankle range of motion will be assessed at clinic visit. No stretching exercises with the device, but will be provided standard care through physiotherapist in acute cases, and no stretching exercises for chronic patients. Reassessment will be done at six weeks and 10 weeks.
Arm/Group | Standard of Care or Ankle Exerciser
Number analyzed (Participants) | 26
Age, Customized [Count of Participants; unit: Participants]
  18 years or older | 26
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male and Female | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Range of Motion
Description: Participants randomized into ARM stretching device group will experience less ankle stiffness and an increased range of motion after using the stretching device, as compared to the control group receiving traditional physiotherapy.
Time Frame: Ten weeks
Population: No participant data or results are available as the investigator left the institution without making them or any analysis available.
Groups:
- Standard of Care: Patient ankle range of motion will be assessed at clinic visit. No stretching exercises with the device, but will be provided standard care through physiotherapist in acute cases, and no stretching exercises for chronic patients. Reassessment will be done at six weeks and 10 weeks.Patient ankle range of motion will be assessed at clinic visit. They will either receive standard care physiotherapy, or use the ankle exerciser in the following manner:
  Subjects will train using only one combination of movement, dorsiflexion with inversion. This is done by manipulating the ring so that the medial and anterior ropes are taut. Subject will start with 3 minute warm-up. Subject will then manipulate the ring so that the foot moves into dorsiflexion with inversion until a point of tolerable discomfort is felt; subject will hold this position for 30 seconds. Stretch will be repeated 10 times, each day, for six weeks.
  Reassessment will be done at six weeks and 10 weeks.
Arm/Group | Standard of Care
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 10 weeks
Description: Adverse event information not available as investigator left the institution without providing this information or making it available.
Groups:
- Standard of Care or Ankle Exerciser: Patient ankle range of motion will be assessed at clinic visit. No stretching exercises with the device, but will be provided standard care through physiotherapist in acute cases, and no stretching exercises for chronic patients. Reassessment will be done at six weeks and 10 weeks.Patient ankle range of motion will be assessed at clinic visit. They will either receive standard care physiotherapy, or use the ankle exerciser in the following manner:
  Subjects will train using only one combination of movement, dorsiflexion with inversion. This is done by manipulating the ring so that the medial and anterior ropes are taut. Subject will start with 3 minute warm-up. Subject will then manipulate the ring so that the foot moves into dorsiflexion with inversion until a point of tolerable discomfort is felt; subject will hold this position for 30 seconds. Stretch will be repeated 10 times, each day, for six weeks.
  Reassessment will be done at six weeks and 10 weeks.
Arm/Group | Standard of Care or Ankle Exerciser
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
No participant data were analyzed because the investigator left the institution before doing so. The results are unavailable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes